CLINICAL TRIAL: NCT01357772
Title: Randomized Placebo-controlled Phase III Trial of Low Dose Tamoxifen in Women With Breast Intraepithelial Neoplasia - Long Term Follow-up
Brief Title: Trial of Low Dose Tamoxifen in Women With Breast Intraepithelial Neoplasia - Long Term Follow-up
Acronym: TAM-01
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Andrea DeCensi (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other); European Institute of Oncology (Other)
Responsible Party: Sponsor-Investigator, Andrea DeCensi, Medical Oncology Director, Ente Ospedaliero Ospedali Galliera
Organization: Ente Ospedaliero Ospedali Galliera (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GAL 01; 2007-007740-10 (EudraCT Number)
Record Dates: First submitted 2011-05-17; First posted 2011-05-23 (Estimated); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Carcinoma, Intraductal, Noninfiltrating; Recurrence, Local Neoplasm; Breast Neoplasms; Atypical Hyperplasia
Keywords: DCIS; tamoxifen; dose reduction
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Neoplasm Recurrence, Local; Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tamoxifen (Experimental): tamoxifen at daily dose of 5 mg for a total treatment time of 3 years
  Interventions: Drug: Tamoxifen
- placebo (Placebo Comparator): placebo at daily dose of 5 mg for a total treatment time of 3 years
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Tamoxifen
  Other Names: Tamoxifen citrate (ATC code: L02BA01)
  Arms: Tamoxifen
Drug: placebo
  Arms: placebo

SUMMARY:
The aim of the study is to evaluate whether tamoxifen at a low dose of 5mg/d reduces in the long term the incidence of invasive breast cancer and ductal carcinoma in situ, DCIS (DIN 1c, 2, 3) of the breast, in woman operated for lobular intraepithelial neoplasia (LIN1, 2 and 3) or ER-positive ductal intraepithelial neoplasia (DIN 1b, DIN2, DIN3, 1a excluded) of the breast.

To improve the risk-benefit ratio, the use of lower doses of the drug has been proposed.

Biomarker trials revealed that 5 mg/d was noninferior to 20 mg/d in inhibiting proliferation of breast cancer and normal endometrial tissue.

By contrast, the risk of endometrial cancer si dose-dependent, and the dose reduction can lead a substantial decrease. Morover a dose of 5 mg/day is associated with an overall decrease of the estrogenic activity of tamoxifen on insulin like growth factor (IGF-I), sex hormone-binding globulin (SHBG) and antithrombin-III, with a decrease of venous thromboembolic events. Moreover, tamoxifen exhibits a high tissue distribution, so that a dose of 5 mg/day attains at the breast tissue level a concentration 10 times higher than that needed to inhibit cell growth in vitro.

A prospective cohort study also showed that 10 mg on alternate days halves recurrence of DCIS in postmenopausal women.

It has been shown that the treatment of dysplasia or pre-cancer drives the reduction of the invasive neoplasms onset. This is a chemoprevention trial designed to validatate the low-dose Tamoxifen in women with diseases at high evolutionary risk. The demonstration of efficacy and safety of such a treatment for the prevention of the invasive breast cancer would lead improvements in term of survival and quality of life for the patients at increased risk.

DETAILED DESCRIPTION:
Italian, multicenter, phase III trial: controlled, parallel group comparision, randomized (1:1) duble blind, tamoxifen 5 mg/d versus placebo administered for 3 years. A total of 500 women 75 years of age or younger with newly diagnosed non-invasive breast cancer have been included in the study. The long-term study implies a minimum 10 year follow up after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

1. Women of age ≥ 18 and < 75 years
2. Women operated on for lobular (LIN 2 and 3) or ER positive or unknown ductal DCIS, i.e DIN 1-3, but DIN 1a excluded) intraepithelial neoplasia in the 5 years (60 months) prior the inclusion in the study. Both incident (diagnosis < 12 months) and prevalent cases diagnosis ≥12, and < 60 months) will be included, including recurrent cases
3. ECOG Performance status ≤ 1
4. Written informed consent

Exclusion Criteria:

1. Any type of malignancy, with the exclusion of non-melanoma skin cancer
2. Proliferative disorders of the endometrium such as atypical hyperplasia, endometriosis, unresected polyps, symptomatic myoma
3. Liver, kidney and heart function impairment grade ≥ 2 (CTCAE criteria v.3.0)
4. Any type of retinal disorders, severe cataract and glaucoma
5. Presence of significant risk factors for venous events, including immobilization after trauma within the last 3 months for longer than 2 weeks, deep venous thrombophlebitis or other significant venous thrombotic event,VTE (pulmonary embolism, stroke, etc.)
6. Use of tamoxifen, raloxifene or other selective estrogen receptor modulator (SERMs)
7. Use of anastrozole and other aromatase inhibitors (AI) in the last 12 months for ≥ 6 months
8. Dicoumarol anticoagulant therapy in progress
9. Active infections
10. Severe psychiatric disorders or inability to comply to the protocol procedures
11. Geographic inaccessibility or difficulties in ensuring adequate compliance
12. Women who are pregnant or breastfeeding
13. Any other factor which, at the discretion of the investigator, may controindicate the use of tamoxifen

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2008-11-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of invasive breast cancer events and DCIS | 20 years
  Number of neoplastic events, i.e., invasive breast cancer or ductal carcinoma in situ of the breast from the start of treatment up to at least 16 years from treatment initiation.

SECONDARY OUTCOMES:
Number of other non-invasive breast events | 20 years
  Number of other non-invasive breast disorders (LCIS, atypical ductal or lobular hyperplasia), endometrial cancer, ovarian cancer, thromboembolic events; bone fractures, cardiovascular and thromboembolic events, clinically manifested cataracts and melanoma; change of mammographic density from the start of treatment up to at least 16 years from treatment initiation.
Metabolites of tamoxifen and hormone blood level (in a subgroup of women) | 20 years
  Blood concentrations of metabolites including circulating IGF-I,IGFBP-3, SHBG, hormones (testosterone, estradiol, SHBG, CRP), tamoxifen metabolites (4OH tamoxifen and endoxifen).
CYP2D6 polymorphisms analysis | 20 years
  Esploratory analisis of some SNPS of the cytochrome P450 genes involved in tamoxifen metabolism such as CYP2D6.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea DeCensi, MD, Principal Investigator — E.O.Ospedali Galliera
Locations (14):
- Italy (14):
  - Ospedali riuniti ASL AL - Ospedale SS. Antonio e Margherita, Tortona, Alessandria
  - Istituto Scientifico Romagnolo per lo studio e la cura dei tumori, Meldola, Forlì-Cesena
  - Ospedale di Carpi "Bernardino Ramazzini", Carpi, Modena
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Azienda Ospedaliera Mater Domini Catanzaro, Catanzaro
  - E.O. Ospedali Galliera, Genoa
  - IEO - European Institute of Oncology IRCCS, Milan
  - Azienda Ospedaliera-Universitaria Policlinico di Modena, Modena
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - ICS Maugeri -Centro Medico di Pavia, Pavia
  - AUSL - Oncologia Medica, Ravenna
  - Azienda Ospedaliera-Universitaria Città della Salute e della Scienza di Torino, Torino
  - Azienda Socio-Sanitaria Territoriale Sette Laghi, Varese, Varese
  - Azienda ULSS8 Berica, Vicenza

IPD SHARING:
Plan to Share IPD: Yes
Authors are open to share data based on a request for collaboration that includes a data analysis plan.
  Please send an e-mail to both: andrea.decensi@galliera.it; mpuntoni@ao.pr.it
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Result] DeCensi A, Puntoni M, Johansson H, Guerrieri-Gonzaga A, Caviglia S, Avino F, Cortesi L, Ponti A, Pacquola MG, Falcini F, Gulisano M, Digennaro M, Cariello A, Cagossi K, Pinotti G, Lazzeroni M, Serrano D, Briata IM, Buttiron Webber T, Boni L, Bonanni B. Effect Modifiers of Low-Dose Tamoxifen in a Randomized Trial in Breast Noninvasive Disease. Clin Cancer Res. 2021 Jul 1;27(13):3576-3583. doi: 10.1158/1078-0432.CCR-20-4213. Epub 2021 Feb 19. PMID 33608319
- [Result] Lazzeroni M, Serrano D, Dunn BK, Heckman-Stoddard BM, Lee O, Khan S, Decensi A. Oral low dose and topical tamoxifen for breast cancer prevention: modern approaches for an old drug. Breast Cancer Res. 2012 Oct 29;14(5):214. doi: 10.1186/bcr3233. PMID 23106852
- [Result] DeCensi A, Johansson H, Helland T, Puntoni M, Macis D, Aristarco V, Caviglia S, Webber TB, Briata IM, D'Amico M, Serrano D, Guerrieri-Gonzaga A, Bifulco E, Hustad S, Soiland H, Boni L, Bonanni B, Mellgren G. Association of CYP2D6 genotype and tamoxifen metabolites with breast cancer recurrence in a low-dose trial. NPJ Breast Cancer. 2021 Mar 25;7(1):34. doi: 10.1038/s41523-021-00236-6. PMID 33767162
- [Result] Lazzeroni M, Puntoni M, Guerrieri-Gonzaga A, Serrano D, Boni L, Buttiron Webber T, Fava M, Briata IM, Giordano L, Digennaro M, Cortesi L, Falcini F, Serra P, Avino F, Millo F, Cagossi K, Gallerani E, De Simone A, Cariello A, Aprile G, Renne M, Bonanni B, DeCensi A. Randomized Placebo Controlled Trial of Low-Dose Tamoxifen to Prevent Recurrence in Breast Noninvasive Neoplasia: A 10-Year Follow-Up of TAM-01 Study. J Clin Oncol. 2023 Jun 10;41(17):3116-3121. doi: 10.1200/JCO.22.02900. Epub 2023 Mar 14. PMID 36917758
- [Derived] Carbone A, Oliva M, Puntoni M, Guerrieri-Gonzaga A, Briata IM, Lazzeroni M, Serrano D, Giordano L, Digennaro M, Cortesi L, Millo F, Cagossi K, Aprile G, Serra P, Gallerani E, Bonanni B, DeCensi A. Effect of low-dose tamoxifen on benign gynecological and breast conditions in a phase III trial in non-invasive breast cancer. J Natl Cancer Inst. 2025 Aug 28:djaf250. doi: 10.1093/jnci/djaf250. Online ahead of print. PMID 40880294
- [Derived] DeCensi A, Puntoni M, Guerrieri-Gonzaga A, Caviglia S, Avino F, Cortesi L, Taverniti C, Pacquola MG, Falcini F, Gulisano M, Digennaro M, Cariello A, Cagossi K, Pinotti G, Lazzeroni M, Serrano D, Branchi D, Campora S, Petrera M, Buttiron Webber T, Boni L, Bonanni B. Randomized Placebo Controlled Trial of Low-Dose Tamoxifen to Prevent Local and Contralateral Recurrence in Breast Intraepithelial Neoplasia. J Clin Oncol. 2019 Jul 1;37(19):1629-1637. doi: 10.1200/JCO.18.01779. Epub 2019 Apr 11. PMID 30973790
- See also: PubMed ID: 33608319 — https://pubmed.ncbi.nlm.nih.gov/33608319/
- See also: PubMed ID: 23106852 — https://pubmed.ncbi.nlm.nih.gov/23106852/
- See also: PubMed ID: 33767162 — https://pubmed.ncbi.nlm.nih.gov/33767162/
- See also: PMID: 36917758 — https://pubmed.ncbi.nlm.nih.gov/36917758/